CLINICAL TRIAL: NCT02779205
Title: Evaluation of Tissue Regeneration Potential (in the Skin) of Child's Adipose Cells During the Development.
Brief Title: Child's Adipose Cells: Capacity of Tissue Regeneration
Acronym: cicASChild
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11 228 02; 2011-A01469-32 (Registry Identifier: Agence National du Médicament et des Produits de santé)
Record Dates: First submitted 2015-07-10; First posted 2016-05-20 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Burns
Keywords: Cell therapy; Stromal Cells; Stem cells; Adipose tissue; Children
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0-1 year old child (Other): Adipose tissue sample in 0-1 year old child with an act of surgery settled by cure of inguinal hernia, or by vesico-ureteral ebb by abdominal way
  Interventions: Procedure: adipose tissue sample
- >1-10 year old child (Other): Adipose tissue sample in >1-10 year old child with an act of surgery settled by cure of inguinal hernia, or by vesico-ureteral ebb by abdominal way
  Interventions: Procedure: adipose tissue sample

INTERVENTIONS:
Procedure: adipose tissue sample — adipose tissue sample

SUMMARY:
The beneficial effect related to the administration of adipose tissue-derived stromal cells (ADSC) is demonstrated in various situations of physiological and pathological wound healing, thus opening a new field for cell therapy. Despite the use of new technologies, management of burns in children as well as congenital malformation such as hypospadias and cleft lip and/ or cleft palate can lead to aesthetic and functional sequelae requiring multiple surgical procedures. Cell therapy based on the administration of the ADSC seems a promising issue in such indications, however, to date no study has been conducted with ADSC from a pediatric population. An initial study (Protocol 0808203) allowed investigors to obtain the first samples of adipose tissue from children and to conduct an in vitro comparative study on the characterization and properties of the ADSC from children compared to adults. In the continuity, this second study aims to complete knowledge on the efficacy and safety of children ADSC cell therapy assessed in an animal model of skin wound healing developed in the lab.

DETAILED DESCRIPTION:
Through this study, the medium term objective is to approach a clinical protocol for treatment of pathological scars in developing an appropriate way to deliver ADSC for a future clinical application, while ensuring the safety of such procedure.

The primary goal of this work is to determine whether ADSC from children prepared according to Good Manufacturing Practice (GMP), is associated with an improvement of wound healing in vivo as demonstrated with adult ADSC. To answer this question, 40 samples of adipose tissue of children obtained from settled surgery (inguinal hernia and vesico-ureteral reflux by suprapubic way) will be performed within the 2 groups of children; 0 to 1 year and 2 to 13 years, defined from data acquired in the previous protocol. Wound healing will be evaluated in a nude mouse model of skin burn. A macroscopic analysis will be carried out with two indexes described in the literature (re-epithelialization and scar contraction) and expressed as a percentage of the initial lesion at different times (3 days, 7 days, 10 days, 14 days, 21 days, 30 days). A microscopic analysis will be conducted to determine the rate of re-epithelialization (day 7) and the evolution of the skin structural parameters (dermal and epidermal thickness, density of collagen, inflammatory infiltration). These indexes will be defined in the treated group (burned mice and injected with pediatric ADSC) from control mice (burned but not injected with cells). A comparative analysis between the two groups of age will be conducted that will be also compared to data collected with adult ADSC.

To answer to the second part of this primary goal regarding to safety, the study will perform a long-term follow-up (1 yr) of burned mice injected with of ADSC, to obtain data in the animal after transplantation of cells and for further clinical study.

Complementary in vitro investigations still seems necessary to better understand the specificities of ADSC from pediatric origin and particularly to perform transcriptomic and epigenetic studies.

ELIGIBILITY:
INCLUSION CRITERIA:

* absence of tumor pathology, known systemic or chronic viral
* absence of long-term treatment
* signing informed consent form of persons exercising parental authority

  1st group (20 children):
* Between 0 and less than or equal to 1 year
* Weighing at least 1500 g at birth
* Age ≥ 37 weeks of amenorrhea

  2nd group (20 children)
* Older than 1 year to 10 years

EXCLUSION CRITERIA:

* Children whose age is above 10 years
* premature babies with birth weight under 1500 grams
* Any child with a tumor pathology, a systemic disease, or whose serology (viral) would be known as positive (HIV 1 and 2, hepatitis B, C, ...).
* Any child following a long term treatment.

Ages: 37 Weeks to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Efficacity of treatment as assessed by surface healed skin (cm2) in animal model | 1 month after injection
  Efficacy of ADSC in animal model healing
Efficacity of treatment as assessed by surface healed skin (cm2) in animal model | 1 year after injection
  Efficacy of ADSC in animal model healing
Security as assessed by absence of tumorigenicity at injection site in animal model | 1 month after injection
  Clinical security of treatment
Security as assessed by absence of tumorigenicity at injection site in animal model | 1 year after injection
  Clinical security of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GALINIER, MD, PhD, Principal Investigator — Chirurgie pédiatrique - Hôpital des enfants
Locations (1):
- CHU de Toulouse-Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbo O, Taurand M, Monsarrat P, Raymond I, Arnaud E, De Barros S, Auriol F, Galinier P, Casteilla L, Planat-Benard V. Comparison between pediatric and adult adipose mesenchymal stromal cells. Cytotherapy. 2017 Mar;19(3):395-407. doi: 10.1016/j.jcyt.2016.11.012. Epub 2016 Dec 28. PMID 28040462